CLINICAL TRIAL: NCT07024589
Title: A Phase 1, Single-Center, Randomized, Blinded, Placebo-Controlled Trial in Healthy Adults to Evaluate the Safety, Tolerability, and Pharmacokinetics of Single and Multiple Doses of Oral AN2-502998
Brief Title: First-in-Human Trial of Oral AN2-502998
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: AN2 Therapeutics, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Basic Science
Other Study IDs: 998-101
Record Dates: First submitted 2025-05-31; First posted 2025-06-17 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Healthy Volunteers
Keywords: AN15368; AN2-502998; AN2 Therapeutics; Benzoxaborole; Boron; Chagas disease; Healthy Volunteer; Phase 1; Trypanosoma cruzi; T. cruzi
MeSH Terms: conditions — Chagas Disease

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Single Ascending Dose (SAD) (Experimental): Participants will be randomized in a 3:1 ratio to receive a single dose of either AN2-502998 or placebo.
  Interventions: Drug: AN2-502998; Drug: Placebo
- Multiple Ascending Dose (MAD) (Experimental): Participants will be randomized in a 3:1 ratio to receive multiple doses of either AN2-502998 or placebo.
  Interventions: Drug: AN2-502998; Drug: Placebo

INTERVENTIONS:
Drug: AN2-502998 — Oral Capsule
Drug: Placebo — Oral Capsule

SUMMARY:
First-in-Human Phase 1, Single-Center, Randomized, Blinded, Placebo-Controlled Trial in Healthy Adults to Evaluate the Safety, Tolerability, and Pharmacokinetics of Single and Multiple Doses of Oral AN2-502998

DETAILED DESCRIPTION:
First-in-human Phase 1, Single-Center, Randomized, Blinded, Placebo-Controlled Trial in Healthy Adults to Evaluate the Safety, Tolerability, and Pharmacokinetics of Single and Multiple Doses of Oral AN2-502998

Part A (SAD; Groups SAD1-SAD6):

Part A is the Single Ascending Dose (SAD) portion of the trial that will be conducted in approximately 48 healthy adults in approximately 6 groups. Eight participants in each group will be randomized in a 6:2 ratio to receive a single dose of AN2-502998 or matching PBO, respectively (6 AN2-502998:2 PBO).

Part B (MAD; Groups MAD1-MAD3):

Part B is the Multiple Ascending Dose (MAD) portion of the trial that will be conducted in approximately 24 healthy adults in approximately 3 groups. Eight participants in each group will be randomized in a 6:2 ratio to receive multiple doses of AN2-502998 or matching PBO (6 AN2 502998:2 PBO) QD for 10 days.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female aged 18 to 55 years, inclusive, at Screening
2. Willing and able to provide written informed consent
3. Willing and able to comply with all trial assessments and adhere to the protocol schedule
4. BMI between ≥18 and <32 kg/m2 (inclusive); BMI is calculated as weight measured in kilograms (kg) divided by the square of height measured in meters (m)
5. If female, must:

   1. Be of nonchildbearing potential defined as either postmenopausal for ≥2 years or surgically sterile (bilateral salpingectomy, bilateral oophorectomy, or hysterectomy); postmenopausal is defined as amenorrheic for ≥1 year in the absence of other biological causes, age appropriate, and has a FSH level during Screening indicating a postmenopausal state; AND
   2. Have negative results for pregnancy tests performed as follows:

   i. Urine specimen obtained during Screening, and ii. Serum specimen obtained on Study Day -1
6. If male and sexually active with a female of childbearing potential, must be surgically sterile or agree to practice at least 1 of the following effective forms of contraception up to 90 days after the last dose of study drug, starting with Study Day 1:

   1. Partner(s) using an IUD
   2. Partner(s) using oral, injected, or implanted methods of hormonal contraceptives
   3. Partner(s) with bilateral tubal occlusion
   4. Total abstinence from sexual intercourse as the preferred lifestyle of the participant; periodic abstinence is not acceptable
7. If male, must agree to use a male condom during intercourse to avoid potential drug exposure to the partner up to 90 days after the last dose of study drug, starting with Study Day 1
8. If female, must agree to use a male condom during heterosexual intercourse to avoid potential drug exposure to the partner up to 90 days after the last dose of study drug, starting with Study Day 1
9. Agree to not donate sperm (males) or ova (females) from Screening until 90 days after the last dose of study drug
10. Medically healthy with no significant clinical medical history, physical examination findings, laboratory results, vital signs, or 12-lead ECG findings, as deemed by the Investigator (or delegate)

Exclusion Criteria:

1. History of significant sensitivity to any drug, including any excipients used in AN2-502998
2. Requirement for any over-the-counter and/or prescription medication, vitamins and/or herbal supplements
3. Use of any medications (prescription or over-the-counter), vitamins, and/or herbal supplements within the 2-week period prior to the first dose of study drug administration or within 5 half-lives of the respective medication, whichever is longer
4. Receipt of any drug by injection, including vaccinations, within 30 days (for vaccinations) or a period defined by 5 half-lives, whichever is longer, prior to study drug administration
5. If female, is pregnant or breastfeeding
6. Positive test result for HBsAg, HCV Ab, HIV Ab, or HIV Ag at Screening; negative HIV status will be confirmed at Screening
7. ALT, AST, or total bilirubin with direct bilirubin >ULN for the reference laboratory at Screening
8. CrCl (Cockcroft-Gault formula), Hgb, Hct, WBC, neutrophil, or platelet count <LLN for the reference laboratory at Screening, unless deemed not CS by the Investigator
9. Fasting glucose ≥5.6 mmol/L
10. QTcF interval duration >450 msec for females or >430 msec for males at Screening
11. Recent (3-month) history of drug or alcohol abuse that could preclude adherence to the protocol
12. History of regular alcohol consumption exceeding 7 drinks/week for females or 14 drinks/week for males (1 drink = 5 ounces [150 mL] of wine or 12 ounces [360 mL] of beer, or 1.5 ounces [45 mL] of hard liquor) within 6 months prior to Screening
13. Positive screen for drugs of abuse, alcohol, or cotinine at Screening and Study Day -1
14. History of seizures, diabetes, or cancer (except basal cell carcinoma of the skin)
15. Current clinically significant cardiovascular, respiratory (except mild asthma), renal, hepatic, gastrointestinal, hematologic, neurologic or thyroid disease, or any uncontrolled medical illness or psychiatric disease or disorder
16. Past history of epilepsy; any clinically significant cardiovascular, respiratory (except mild asthma), renal, hepatic, gastrointestinal, hematologic, neurologic, or thyroid disease; or any uncontrolled medical illness or psychiatric disease or disorder
17. History of gastric surgery, vagotomy, bowel resection, cholecystectomy, or any surgical procedure or medical condition that might interfere with gastrointestinal motility, pH, or absorption
18. Donation or loss of 550 mL or more blood volume (including plasmapheresis) within 4 weeks prior to study drug administration or receipt of a transfusion of any blood product within 8 weeks prior to study drug administration
19. Receipt of any investigational product within a period equal to 10 half-lives of the product, if known, or a minimum of 6 weeks prior to study drug administration
20. Consumption of alcohol within the 72 hours prior to study drug administration
21. Consumption of grapefruit, star fruit, Seville oranges, or products containing any of these ingredients within the 10-day period prior to study drug administration
22. Use of inhaled nicotine, tobacco, or marijuana products within the 6 months prior to study drug administration
23. Current enrollment in another clinical trial

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 72 (Estimated)
Dates: Start 2025-08-04 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Evaluate the Incidence of Treatment Emergent Adverse Events at Baseline and Through Study Completion for a Single Dose | Day 1 through last follow-up (9 Days after single dose)
  Incidence, relatedness, and severity of adverse events
Evaluate Physical Examination Abnormalities from Baseline Through Study Completion for a Single Dose | Day 1 through last follow-up (9 Days after single dose)
  Incidence of physical exam abnormalities
Evaluate Change in Vital Signs from Baseline Through Study Completion for a Single Dose | Day 1 through last follow-up (9 Days after single dose)
  Incidence of changes in blood pressure, pulse, respiratory rate, and temperature
Evaluate Changes in 12-lead ECG Measurements from Baseline Through Study Completion for a Single Dose | Day 1 through last follow-up (9 Days after single dose)
  Incidence of changes in 12-lead ECG parameters from baseline
Evaluate Changes in Clinical Laboratory Tests from Baseline Through Study Completion for a Single Dose | Day 1 through last follow-up (9 Days after single dose)
  Incidence of changes in clinical laboratory measurements from baseline
Evaluate the Incidence of Treatment Emergent Adverse Events at Baseline and Through Study Completion for Multiple Doses | Day 1 through last follow-up (10 Days after last dose)
  Incidence, relatedness, and severity of adverse events
Evaluate Physical Examination Abnormalities from Baseline Through Study Completion for Multiple Doses | Day 1 through last follow-up (10 Days after last dose)
  Incidence of physical exam abnormalities
Evaluate Change in Vital Signs from Baseline Through Study Completion for Multiple Doses | Day 1 through last follow-up (10 Days after last dose)
  Incidence of changes in blood pressure, pulse, respiratory rate, and temperature
Evaluate Changes in 12-lead ECG Measurements from Baseline Through Study Completion for Multiple Doses | Day 1 through last follow-up (10 Days after last dose)
  Incidence of changes in 12-lead ECG parameters from baseline
Evaluate Changes in Clinical Laboratory Tests from Baseline Through Study Completion for Multiple Doses | Day 1 through last follow-up (10 Days after last dose)
  Incidence of changes in clinical laboratory measurements from baseline
Characterize the PK Profile of AN2-502998: Maximum Plasma Concentration | Day 1 through last follow-up (3 Days after last dose)
  Determination of the maximum plasma concentration (Cmax)
Characterize the PK Profile of AN2-502998: Time to Maximum Plasma Concentration | Day 1 through 3 days after last dose
  Determination the time to maximum plasma concentration (Tmax)
Characterize the PK Profile of AN2-502998: Terminal Half-Life | Day 1 through 3 days after last dose
  Determine the apparent terminal half-life (t½)
Characterize the PK Profile of AN2-502998: Area Under Plasma Concentration Curve | Day 1 through 3 days after last dose
  Area under plasma concentration-time curve from zero to a designated dosing interval
Characterize the PK Profile of AN2-502998: Apparent Plasma Clearance | Day 1 through 3 days after last dose
  Apparent plasma clearance of drug after extravascular administration CL/F

CONTACTS AND LOCATIONS:
Locations (1):
- Nucleus Network, Melbourne, Victoria, Australia

IPD SHARING:
Plan to Share IPD: No